CLINICAL TRIAL: NCT04076046
Title: Multicentric Prospective Validation of the Zurich Pituitary Score
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Carlo Serra, Principal investigator, University of Zurich
Other Study IDs: ZPS prospective validation
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pituitary Adenoma
Keywords: pituitary adenoma endoscopic surgery zurich pituitary score
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Predictive analytics for GTR, EOR and RV are useful in surgical decision-making, particularly whenever there is no unequivocal indication for surgery. Several factors have been shown to have a role in predicting GTR. Among these, the Knosp classification has proven over the years to be a good predictor of GTR. The score is based on the lateral extension of the adenoma in relation the the intracranial bedding of the internal carotid artery. However, recent literature has demonstrated that the Knosp classification suffers from relatively poor interrater agreement. Moreover the classification was conceived in an era when endoscopic techniques were not available: nowadays endoscopic technique allows visualization and possibly also reaching portions of adenoma which at the time when the Knosp classification was introduced were simply not possible. Lastly, the efficacy of the Knosp's score in predicting also EOR and RV has never been tested.

Recently a new score - the Zurich Pituitary Score (ZPS) has been proposed at the University Hospital of Zürich (USZ). The score has proved in the examined series to be more powerful than the Knosp classification in predicting GTR, EOR and RV. A good interrater agreement was also demonstrated. The score however, has been validated only in a monocentric setting with a limited number of patients. The aim of this study is to assess the (1) predictive ability of the ZPS for GTR, EOR, and RV, and (2) the inter-rater agreement of the ZPS in an external validation study.

DETAILED DESCRIPTION:
In transsphenoidal surgery (TSS) for pituitary adenoma (PA), gross total resection (GTR) is often the target since it has been shown to relevantly influence long term patient outcome. This applies both to functioning adenomas (FA) as well as to non-functioning adenomas (NFPA). Mounting evidence shows that in cases where GTR is not achievable, maximizing extent of resection (EOR) is still highly desirable, particularly in case of FA, with the aim of obtaining the smallest possible residual volume (RV).

Predictive analytics for GTR, EOR and RV are useful in surgical decision-making, particularly whenever there is no unequivocal indication for surgery. Several factors have been shown to have a role in predicting GTR. Among these, the Knosp classification has proven over the years to be a good predictor of GTR. The score is based on the lateral extension of the adenoma in relation the the intracranial bedding of the internal carotid artery. However, recent literature has demonstrated that the Knosp classification suffers from relatively poor interrater agreement. Moreover the classification was conceived in an era when endoscopic techniques were not available: nowadays endoscopic technique allows visualization and possibly also reaching portions of adenoma which at the time when the Knosp classification was introduced were simply not possible. Lastly, the efficacy of the Knosp's score in predicting also EOR and RV has never been tested.

Recently a new score - the Zurich Pituitary Score (ZPS) has been proposed at the University Hospital of Zürich (USZ). The score has proved in the examined series to be more powerful than the Knosp classification in predicting GTR, EOR and RV. A good interrater agreement was also demonstrated. The score however, has been validated only in a monocentric setting with a limited number of patients. The aim of this study is to assess the (1) predictive ability of the ZPS for GTR, EOR, and RV, and (2) the inter-rater agreement of the ZPS in an external validation study.

ELIGIBILITY:
Inclusion Criteria:

* Patients harboring suspected pituitary adenoma.
* Patients undergoing endoscopic transsphenoidal surgery
* Preoperative MRI including at least one volumetric sequence (i.e. MPRAGE or SPGR) with gadolinium with possibility for coronal reconstructions
* Postoperative MRI (2-4 months postoperative) including at least one volumetric sequence (i.e. MPRAGE or SPGR) with Gadolinium with possibility for coronal reconstructions

Exclusion Criteria:

* Patients undergoing combined or transcranial operations
* Patients for whom a biopsy only is planned
* Patients by whom histology does not confirm the diagnosis of pituitary adenoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive serie of patients undergoing endoscopic transsphenoidal pituitary adenoma surgery
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Gross Total Resection | 2 to 4 months postoperatively
  Gross Total Resection on magnetic resonance imaging
Extent of Resection | 2 to 4 months postoperatively
  Percentage of removed adenoma volume on magnetic resonance imaging
Residual Adenoma Volume | 2 to 4 months postoperatively
  Percentage of original adenoma volume still visible at the postoperative magnetic resonance imaging
Zurich Pituitary Score | On preoperative MRI
  Four-tier score as follows:
  Grade Criteria I R < 0.75 II 0.75 < R < 1.25 III 1.25 < R IV Encasement of the intracavernous ICA
  R = ratio of maximum horizontal tumor diameter divided by the minimum intercarotid distance at the intracavernous horizontal C4 segment of the ICA.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Serra, MD, Study Director — Klinik für Neurochirurgie, UniversitätsSpital Zürich, Switzerland
Locations (10):
- Donald and Barbara Zucker School of Medicine at Hofstra/Northwell, New York, New York, United States
- Department of Neurosurgery, Kepler Universitäts Klinikum, Linz, Austria
- Toronto Western Hospital, University of Toronto, Toronto, Canada
- Department of Neurosurgery and Neurooncology, First Faculty of Medicine, Charles University and Military University Hospital, Prague, Czechia
- Italy (4):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Universita' degli Studi Federico II, Napoli
  - Reparto di Neurochirurgia, Ospedale di Circolo e Fondazione Macchi, Universita' dell'Insubria, Varese
- Switzerland (2):
  - CHUV, Lausanne
  - Department of Neurosurgery, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staartjes VE, Serra C, Maldaner N, Muscas G, Tschopp O, Soyka MB, Holzmann D, Regli L. The Zurich Pituitary Score predicts utility of intraoperative high-field magnetic resonance imaging in transsphenoidal pituitary adenoma surgery. Acta Neurochir (Wien). 2019 Oct;161(10):2107-2115. doi: 10.1007/s00701-019-04018-9. Epub 2019 Aug 7. PMID 31392567
- [Background] Serra C, Staartjes VE, Maldaner N, Muscas G, Akeret K, Holzmann D, Soyka MB, Schmid C, Regli L. Predicting extent of resection in transsphenoidal surgery for pituitary adenoma. Acta Neurochir (Wien). 2018 Nov;160(11):2255-2262. doi: 10.1007/s00701-018-3690-x. Epub 2018 Sep 29. PMID 30267209